CLINICAL TRIAL: NCT05465564
Title: My Hearing Experience - a Study About the Effect of Personality and Lifestyle on Everyday Hearing
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: WSAUD A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: Hear_101
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Hearing Impairment; Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of this study is to investigate how personality, motivation & auditory lifestyle relate to hearing aid satisfaction & acceptance for first-time hearing aid users. As such, first-time hearing aid users will be followed via an app for a period of six months. They will answer baseline questionnaires about personality, lifestyle and hearing aid expectations before the first fit. After the hearing aid fitting, they will be prompted by the app to answer questionnaires about their hearing aid experience at weeks 2, 4, 8, 12, 16, 20 and 24.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years of age
* Sensorineural hearing loss within the hearing aid's fitting range
* Fluency in local language
* First-time hearing aid user
* Experienced smartphone and app user
* Must sign the informed consent

Exclusion Criteria:

* Severe cognitive impairment that would preclude the ability to perform the necessary tasks (as judged by the HCP)
* Inability for the TPs to travel to the clinic during the study period
* Complex hearing disorders such as Ménière's

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First-time hearing aid users
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
overall hearing aid satisfaction | 6 months
  minimum: 1, maximum: 10 ; the higher value indicates a better outcome
IOI-HA | 6 months
  minimum: 7, maximum: 35; the higher value indicates a better outcome
hearing aid satisfaction (Hearing-Related Lifestyle scale) | 6 months
  minimum: 1, maximum: 5; the higher value indicates a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Dina Lelic, Lynge, DK, Denmark